CLINICAL TRIAL: NCT02911974
Title: Randomized Trial Comparing Fine Needle Biopsy and Fine Needle Aspiration Needles for Endoscopic Ultrasound -Guided Sampling of Solid Pancreatic Masses
Brief Title: Comparing Biopsy Needles for Endoscopic Ultrasound Guided Samples for Pancreatic Masses
Acronym: Expect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 889569
Record Dates: First submitted 2016-08-22; First posted 2016-09-23 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Pancreatic Neoplasm
Keywords: fine needle biopsy; EUS; solid pancreatic mass
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acquire EUS Biopsy Device (Active Comparator): All patients will undergo sampling of pancreatic masses using the Acquire EUS Biopsy Device. Both needles will be used, but the needle to be used first will be based on randomization. A minimum of at least one pass and a maximum of 8 passes will be performed using both needle types.
  Interventions: Device: Acquire EUS Biopsy Device
- Expect EUS Aspiration Needle (Active Comparator): All patients will undergo sampling of pancreatic masses using the Expect EUS Aspiration Needle. Both needles will be used, but the needle to be used first will be based on randomization. A minimum of at least one pass and a maximum of 8 passes will be performed using both needle types
  Interventions: Device: Expect EUS Aspiration Needle

INTERVENTIONS:
Device: Acquire EUS Biopsy Device — 1. At EUS, once the pancreatic mass is identified, patients will be randomized to undergo sampling using the 22G Acquire EUS Biopsy Device or Expect EUS Aspiration Needle.
  Arms: Acquire EUS Biopsy Device
Device: Expect EUS Aspiration Needle — 1. At EUS, once the pancreatic mass is identified, patients will be randomized to undergo sampling using the 22G Acquire EUS Biopsy Device or Expect EUS Aspiration Needle.
  Arms: Expect EUS Aspiration Needle

SUMMARY:
This is a randomized prospective clinical study comparing a fine needle biopsy device and an aspiration needle.

DETAILED DESCRIPTION:
At EUS, once the pancreatic mass is identified, patients will be randomized to undergo sampling using the 22G FNA or FNB needle. All patients will undergo sampling of pancreatic masses using both needles but the needle to be used first will be based on randomization. Subsequent passes will be performed by alternate needles and once onsite diagnosis is established using either needle type, more passes will not be performed for onsite diagnostic adequacy. However, a minimum of at least one pass and a maximum of 8 passes will be performed using both needle types. The number of passes needed to achieve diagnostic adequacy using both needles will documented.

Four dedicated passes will then be performed using the initial randomization sequence for cell block. Two passes will be performed using each needle type and the specimen will be preserved in formalin and sent for cell block processing.

If the doctor cannot obtain enough tissue with the study needles, another needle with a different gauge (19 or 25) will be used. This will also be a maximum of 8 passes. Information about the number of needles used, how many passes were performed, any problems with the needles will be collected. If there is not enough tissue available from these passes to establish a diagnosis, the subject will be asked to come back at another time for a repeat procedure.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo EUS
* Patients with solid pancreatic masses on cross-sectional imaging or with jaundice secondary to biliary obstruction
* Able and willing to provide written or verbal consent

Exclusion Criteria:

* Unable to safely undergo EUS for any reason
* Coagulopathy (Prothrombin time > 18 secs, platelet count < 80,000/ml)
* Active alcohol or other drug use or significant psychiatric illness
* Pregnancy
* Unable or unwilling to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-08; Primary Completion 2017-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
The total area of procured tissue between the FNA and FNB needles | 6 months.
  The primary objective of this study is to compare the total area of procured tissue between the FNA and FNB needles in patients undergoing EUS-guided sampling of pancreatic masses.
  Pancreatic masses sampled using the FNB needle should have a tissue area greater than the FNA needle because of the serrated design of the FNB needle tip. This will be measured using a specialized digital image analysis software.
  This hypothesis will be tested by comparing the total tissue area, tumor area within the tissue, stroma area within the tissue, tumor vs. stroma ratio and the macroscopic length of the procured tissue measured in millimeters. The total of these measurements will provide information about the area of procured tissue.

SECONDARY OUTCOMES:
Diagnostic adequacy between the FNA and FNB needles | 6 months
  The secondary objective of this study is to compare the diagnostic adequacy between the FNA and FNB needles in patients undergoing EUS-guided sampling of pancreatic masses.
  Pancreatic masses sampled using the FNB needle should yield diagnostic adequacy with fewer passes as they are expected to procure a greater area tissue than the FNA needle.
  This hypothesis will be tested by comparing the number of passes required to establish a onsite diagnosis using both needle types in individual patients.

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — AdventHealth
Locations (1):
- Center for Interventional Endoscopy - Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hewitt MJ, McPhail MJ, Possamai L, Dhar A, Vlavianos P, Monahan KJ. EUS-guided FNA for diagnosis of solid pancreatic neoplasms: a meta-analysis. Gastrointest Endosc. 2012 Feb;75(2):319-31. doi: 10.1016/j.gie.2011.08.049. PMID 22248600
- [Background] Varadarajulu S, Fraig M, Schmulewitz N, Roberts S, Wildi S, Hawes RH, Hoffman BJ, Wallace MB. Comparison of EUS-guided 19-gauge Trucut needle biopsy with EUS-guided fine-needle aspiration. Endoscopy. 2004 May;36(5):397-401. doi: 10.1055/s-2004-814316. PMID 15100946
- [Background] Bang JY, Hawes R, Varadarajulu S. A meta-analysis comparing ProCore and standard fine-needle aspiration needles for endoscopic ultrasound-guided tissue acquisition. Endoscopy. 2016 Apr;48(4):339-49. doi: 10.1055/s-0034-1393354. Epub 2015 Nov 12. PMID 26561917
- [Result] Ngamruengphong S, Li F, Zhou Y, Chak A, Cooper GS, Das A. EUS and survival in patients with pancreatic cancer: a population-based study. Gastrointest Endosc. 2010 Jul;72(1):78-83, 83.e1-2. doi: 10.1016/j.gie.2010.01.072. PMID 20620274
- [Result] Othman MO, Wallace MB. The role of endoscopic ultrasonography in the diagnosis and management of pancreatic cancer. Gastroenterol Clin North Am. 2012 Mar;41(1):179-88. doi: 10.1016/j.gtc.2011.12.014. Epub 2012 Jan 16. PMID 22341257